CLINICAL TRIAL: NCT00273000
Title: The Importance of Glucagon-Like Peptide-2 (GLP-2)in Mesenteric Bloodflow in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GLP-2, MBF
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-10

CONDITIONS: Healthy

INTERVENTIONS:
Drug: GLP-2

SUMMARY:
The purpose of this study is to study the effect of GLP-2 on mesenteric bloodflow in healthy adults by the use of ultrasound., it is the hypothesis that GLP-2 vil increase the bloodflow.

DETAILED DESCRIPTION:
The investigation will include 10 testpersons.

It will be a 2 fase study over 2 days.

day 1: The testperson will meet fasting, and take in a standard liquid meal, after this the bloodflow in a mesenteric artery will be measured by use of ultrasonic technique. Bloodsamples will be taken regular in a total wolumne of 200 ml.

day 2:The testperson will meet fasting, there wil be administered intraveneous GLP-2 in 3 increasing doses over 3 x 45 min.and one subcutaneous dose. During this the bloodflow in a mesenteric artery will be measured by use of ultrasonic technique. Bloodsamples will be taken regular in a total wolumne of 200 ml.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* use of drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Mads Hornum, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen City, Denmark